CLINICAL TRIAL: NCT00113256
Title: Randomized Trial of Orathecin and Gemcitabine Versus Placebo and Gemcitabine in Patients With Non-Resectable Pancreatic Cancer Who Have Not Already Received Chemotherapy
Brief Title: Orathecin + Gemcitabine Versus Placebo + Gemcitabine in Chemonaive Non-Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-RUB-048
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
Keywords: rubitecan; Orathecin; 9-nitrocamptothecin; gemcitabine; Gemzar; pancreatic cancer; adenocarcinoma; RFS 2000
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — rubitecan

INTERVENTIONS:
Drug: Rubitecan

SUMMARY:
Patients will be treated with gemcitabine and Orathecin (rubitecan) capsules to evaluate the current estimate of overall survival as a study endpoint prior to launching the blinded randomized phase (versus gemcitabine and placebo) of the study. Toxicity of the drug combination will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age.
* The patient has histologically or cytologically confirmed, non-resectable, Stage II-IV primary adenocarcinoma of the pancreas.
* The patient has had a baseline computed tomography (CT) scan, or magnetic resonance imaging (MRI), to evaluate tumor(s) within 28 days prior to randomization.
* The patient has never been treated with prior chemotherapy, with the exception of low-dose 5-fluorouracil (5-FU) as a radiation sensitizer.
* The patient has sufficiently recovered from the effects of previous surgery (no less than 3 weeks prior to randomization), radiotherapy, and/or immunotherapy (no less than 4 weeks prior to randomization).
* The patient's estimated life expectancy is at least 12 weeks.
* The patient has a Karnofsky Performance Status between 50 and 100.
* The patient has adequate bone marrow function.
* The patient has adequate hepatic and renal function.

Exclusion Criteria:

* The patient has any active, uncontrolled infection requiring antibiotics.
* The patient has any serious, uncontrolled concomitant systemic disorder.
* The patient has surgery scheduled within 8 weeks following initiation of treatment.
* The patient is pregnant or nursing.
* The patient is not capable of consistent oral intake of at least 3 L/day of fluid and/or requires constant intravenous (IV) hydration or frequent tube feeding.
* The patient is receiving any investigational agent(s) or has been a participant in a clinical trial within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-02; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
survival

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Compassionate Cancer Care Medical Group, Corona, California
  - 11100 Warner Avenue, Ste. 200, Fountain Valley, California
  - The Cancer Research & Prevention Center, Soquel, California
  - Mile High Oncology, Denver, Colorado
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Oncology, Baton Rouge, Louisiana
  - N. Mississippi Hematology & Oncology Associates, Tupelo, Mississippi
  - Kansas City Cancer Center, Kansas City, Missouri
  - Cancer Research of Long Island, Great Neck, New York
  - Charleston Hematology Oncology, PA, Charleston, South Carolina